CLINICAL TRIAL: NCT06053983
Title: Comparison Between Atorvastatin and Rosuvastatin in Reduction of Inflammatory Biomarkers in Patients With Acute Coronary Syndrome
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Rawalpindi Medical College (Other)
Responsible Party: Principal Investigator, Naima Shehzadi Qazi, Dr. NAIMA SHEHZADI QAZI PGT MD CARDIOLOGY, Rawalpindi Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 46 /IREFIRMU 2021
Record Dates: First submitted 2023-09-19; First posted 2023-09-26 (Actual); Last update posted 2023-10-17 (Actual); Status verified 2023-10

CONDITIONS: Mi Q Wave
MeSH Terms: interventions — Rosuvastatin Calcium; Atorvastatin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- rosuvastatin 20 mg (Experimental)
  Interventions: Device: Turbox CRP kit; Drug: rosuvastatin 20 mg,
- atorvastatin 40 mg (Experimental)
  Interventions: Device: Turbox CRP kit; Drug: atorvastatin 40 mg

INTERVENTIONS:
Device: Turbox CRP kit — Quantitative estimation of hs-CRP will be conducted at the beginning of the study and after the treatment period using the Turbox CRP kit, which employs turbidimetry as the method of measurement.
Drug: rosuvastatin 20 mg, — The statin are most commonly used agents for prevention of cardiovascular events and recurrent episodes of ACS. Apart from their anti-lipid actions, statins show pleotropic effects which include their anti-inflammatory role. Atorvastatin and rosuvastatin are both members of statin family and have showed their effectiveness in reduction of inflammatory biomarkers in addition to their lipid lowering effects
  Arms: rosuvastatin 20 mg
Drug: atorvastatin 40 mg — The statin are most commonly used agents for prevention of cardiovascular events and recurrent episodes of ACS. Apart from their anti-lipid actions, statins show pleotropic effects which include their anti-inflammatory role. Atorvastatin and rosuvastatin are both members of statin family and have showed their effectiveness in reduction of inflammatory biomarkers in addition to their lipid lowering effects
  Arms: atorvastatin 40 mg

SUMMARY:
This study will help us to compare atorvastatin and rosuvastatin in terms of their ability to reduce biomarkers of inflammation in patients of acute coronary syndrome

ELIGIBILITY:
Inclusion Criteria:

1. Patients with age 18 years and above, of both genders, diagnosed with acute coronary syndrome (as per operational definition) who were not taking statins previously.
2. Patients who sign written informed consent to participate in the study.

Exclusion Criteria:

* 1.Patients who are taking either statins and/or any other drug which lower serum lipid levels, patients with a history of statin hypersensitivity, patients in whom statins are contraindicated.

  2.Patients who will be surgically managed will be also excluded. 3.if coronary revascularization will be planned or anticipated at the time of screening.

  4.Pregnant or lactating women. 5.Patients having concomitant infections which cause the rise of inflammatory markers.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 126 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-08-01 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Mean Change C-reactive protein | AFTER 4 WEEKS
  hs -CRP (mg/l)

CONTACTS AND LOCATIONS:
Overall Officials: asma khan, Study Director — Rawalpindi Medical College
Locations (1):
- Rawalpindi Medical University, Rawalpindi, Pakistan

IPD SHARING:
Plan to Share IPD: No